CLINICAL TRIAL: NCT07377617
Title: Effect of Individualized Education and Exercise Program on Foot Health: Randomized Controlled Trial
Brief Title: Individualized Education and Exercise on Foot Health
Acronym: Foot Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Seyda Can, associate professor, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/168
Record Dates: First submitted 2024-11-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Foot Diseases; Education; Nurse
Keywords: individualized education; exercise program; foot health; nurse; physiotherapist
MeSH Terms: conditions — Foot Diseases | interventions — Resistance Training

STUDY DESIGN:
Masking Description: Analysis will be performed by an expert who is not involved in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An individualized education and exercise program (Experimental): An individualized education and exercise program will be applied to the nurses to improve foot health.
  Interventions: Behavioral: individualized education
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Behavioral: individualized education — An individualized education and exercise program will be applied to the nurses to improve foot health.
  Other Names: exercise program
  Arms: An individualized education and exercise program

SUMMARY:
The purpose of the study is to determine the effect of an individualized education and exercise program applied to nurses on the knowledge, skills and habits of employees regarding foot health. This study is a randomized controlled trial.

The universe of the study will be nurses working in a Training and Research Hospital, and the sample will consist of nurses who agree to participate in the study between the specified dates and meet the criteria. It has been determined that a total of 70 people should be included in the study, 35 in the intervention and control groups.

DETAILED DESCRIPTION:
This article will address the following questions:

1. How is the foot health of the nurses according to the "self-foot health assessment scale"?
2. Is the individualized education and exercise program given to nurses effective on the foot health of employees?

The hypotheses of the study are as follows:

H1: The foot health of the experimental group is more positive than the control group.

H1: The satisfaction levels of the experimental group regarding the foot health program are higher than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Wanting to participate in the study voluntarily,
* Being a nurse.

Exclusion Criteria:

* Not wanting to participate in the study,
* Not being a nurse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Performing exercises related to foot health | 6 weeks
  1. Primary Outcome Measure Outcome Measure Title: Change from Baseline in Self-Foot Health Assessment Instrument (S-FHAI) Score at 6 weeks.
  Description: The S-FHAI is a self-assessment tool consisting of 22 items across 4 categories: skin health (11 items), toenail health (5 items), foot structure (5 items), and foot pain (2 items). Items are primarily evaluated using "Yes/No" responses, while the final item regarding pain intensity uses a 5-point Likert scale (0=no pain, 4=worst imaginable pain). The total score is used to assess the individual's foot health status. Higher scores indicate different levels of foot health across the specified domains.
  Time Frame: Baseline and 6 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 01.01.2025-31.12.2025
Access Criteria: The study protocol will be shared with researchers who request it.